CLINICAL TRIAL: NCT01958554
Title: Randomised Controlled Trial of an Integrated Intervention on Mental Health in Survivors of Intimate Partner Violence
Brief Title: Impact of an Integrated Intervention on Mental Health in Survivors of Intimate Partner Violence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Macmillan Research Group UK (Industry)
Collaborators: NMP Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mac/NMP 0917
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Domestic Violence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): The integrated intervention consisted of 12 week of program and group support, based on the freedom program by pet craven. The former component was provided covering beliefs held and tactics used by the domestic violence abusers and took about 45 minutes. It included protection and enhanced choice-making and problem-solving skills.
  Interventions: Behavioral: Intervention Group
- Wait list control group (No Intervention): The group was listed in wait list and were offered the same intervention and support on completion of study period.

INTERVENTIONS:
Behavioral: Intervention Group
  Arms: Intervention Group

SUMMARY:
Intimate partner violence (IPV) against women have negative mental health consequences for survivors; interventions designed to improve survivors' depressive symptoms and health status are limited.Present study evaluate the effectiveness of an integrated intervention in reducing intimate partner violence (IPV) improving health status.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18
* For those who agreed to participate
* Given written consent
* Screening for abuse was positive

Exclusion Criteria:

* Screened Negative
* serious mental condition including suicide, hallucination, Dementia
* Drug or substance abuse, alcoholism
* Pregnant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Depression | Change from Baseline in Beck Depression Inventory at 12 weeks

SECONDARY OUTCOMES:
Health Related Quality of Life | Change from baseline in SF-36 at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bharat Chaudhari, MA, Study Director — Sonal Foundation, India; Neha sharma, PhD, Study Chair — Macmillan Research Group
Locations (1):
- Sonal Foundation, Mahesāna, Gujarat, India